CLINICAL TRIAL: NCT04709562
Title: Hypercapnia Clinical Efficacy by NIPPV v HVNI: A Randomized Control Trial in the Stabilization of Acute Hypercarbic Respiratory Failure
Brief Title: Clinical Stabilization of Hypercapnia: NIPPV v HVNI
Acronym: HYPERACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: Erlanger Baroness Hospital (Other Government); The Cooper Health System (Other); Dignity Health Medical Foundation (Other); George Washington University (Other); Madigan Army Medical Center (U.S. Federal Agency); Valley Presbyterian Hospital (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-VTPF2020001Sci
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hypercapnic Respiratory Failure; Chronic Obstructive Pulmonary Disease; Dyspnea; Hypercapnic Acidosis
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Dyspnea; Acidosis, Respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Velocity Nasal Insufflation (HVNI) (Experimental): Patients randomly assigned to this arm will be placed on HVNI therapy with an appropriately fitted Vapotherm Prosoft HVNI nasal cannula. Physiologic and ventilation parameters will be recorded.
  Interventions: Device: High Velocity Nasal Insufflation (HVNI)
- Noninvasive Positive Pressure Ventilation (NIPPV) (Active Comparator): Patients randomly assigned to this arm will be placed on NIPPV therapy with an appropriately fitted full face mask using a pressure support mechanical ventilator system. Physiologic and ventilation parameters will be recorded.
  Interventions: Device: Noninvasive Positive Pressure Ventilation (NIPPV)

INTERVENTIONS:
Device: High Velocity Nasal Insufflation (HVNI) — The purpose of this intervention is to evaluate the efficacy of HVNI in clinically stabilizing patients presenting with hypercapnic respiratory distress.
  Other Names: Vapotherm Precision Flow Plus
  Arms: High Velocity Nasal Insufflation (HVNI)
Device: Noninvasive Positive Pressure Ventilation (NIPPV) — The purpose of this intervention is to evaluate the efficacy of NIPPV in clinically stabilizing patients presenting with hypercapnic respiratory distress.
  Other Names: Philips Respironics V60
  Arms: Noninvasive Positive Pressure Ventilation (NIPPV)

SUMMARY:
This study will evaluate the ability of High Velocity Nasal Insufflation [HVNI] to effect ventilation and related physiologic responses in hypercapnic patients when compared to noninvasive positive pressure ventilation [NIPPV].

DETAILED DESCRIPTION:
The overall objective of this randomized study is to evaluate the efficacy of HVNI, in comparison to NIPPV, to clinically stabilize and provide respiratory therapy to patients who have COPD with moderate-to-severe hypercapnic respiratory distress upon presentation. It is hypothesized that HVNI is comparable to NIPPV in the stabilization and relief of moderate-to-severe hypercapnic respiratory distress upon presentation, by relieving the patient's dyspnea (breathlessness) within 4 hours to a comparable degree to NIPPV.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older with a known or suspected diagnosis of COPD
* Presentation with acute hypercapnic respiratory failure
* Moderate to Severe patient baseline hypercarbia/hypercapnia, defined as a baseline PCO2 of 60 mmHg or higher
* Venous pH of 7.0 - 7.35

Exclusion Criteria:

* Severe metabolic derangements (e.g. suspected drug overdose, mixed acid/base disorder)
* Need for airway protection
* Primary condition of Congestive Heart Failure
* Need for emergent intubation
* Pneumonia diagnosis with significant infiltrate on chest x-ray that is clinically correlated with pneumonia
* Inability to provide informed consent
* Pregnancy
* Known contraindication to perform procedures listed, or therapies described in the protocol
* Respiratory arrest or significant respiratory depression on presentation
* Significant nasal occlusion either unilateral or bilateral
* Absence of spontaneous respiration or known contraindication to HVNI
* Extreme agitation or uncooperativeness that would hinder either arm of randomized therapy
* Determined by the clinician to be sufficiently unstable or unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Meltzer, MD, MS, Principal Investigator — George Washington University; Christopher W Jones, MD, Principal Investigator — The Cooper Health System; Anthony Innabi, MBA, RRT-NPS, Principal Investigator — Dignity Health Medical Foundation; Joshua Oliver, MD, Principal Investigator — Madigan Army Medical Hospital; Cynthia Pfeiffer, MD, Principal Investigator — Valley Presbyterian Hospital; Richard Wilkerson, MD, Principal Investigator — University of Maryland; David Yamane, MD, Principal Investigator — George Washington University
Locations (7):
- United States (7):
  - Valley Presbyterian Hospital, Los Angeles, California
  - Dignity Health - St. John's Regional Medical Center, Oxnard, California
  - George Washington University Hospital, Washington D.C., District of Columbia
  - University of Maryland, Baltimore, Maryland
  - Cooper University Hospital, Camden, New Jersey
  - Erlanger Health System, Chattanooga, Tennessee
  - Madigan Army Medical Center, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Started | 36 | 32
Completed | 36 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV) | Total
Number analyzed (Participants) | 36 | 32 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years old] | 63.8 (11.18) | 67.7 (9.44) | 65.96 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 20 | 16 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 36 | 32 | 68

OUTCOME MEASURES:

1. Primary Outcome: Rated Perceived Dyspnea [RPD]
Description: Patient's subjective assessment of their dyspnea, rated as a modified Borg score on a scale from 0 to 10. Higher scores indicate a worse outcome.
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: The participants had to have an RPD reading at all four time points.
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
units on a scale (0-10)
  Baseline | 5.4 (2.93) | 5.6 (2.41)
  30 Min: number analyzed (Participants) | 32 | 26
  30 Min | 3.97 (2.82) | 4.54 (1.65)
  60 Min: number analyzed (Participants) | 32 | 26
  60 Min | 3.09 (2.70) | 4.07 (1.77)
  240 Min: number analyzed (Participants) | 32 | 25
  240 Min | 3.17 (2.59) | 3.34 (2.04)

2. Secondary Outcome: Patient Vital Signs - Heart Rate [HR]
Description: Heart rate, measured in beats per minute (bpm)
Time Frame: During four time points in the study; Baseline, 30 min, 60 min, and 240 min
Population: Patients who had their Heart Rate collected during the four time points in the study.
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
BPM
  Baseline | 93.2 (17.37) | 85.9 (16.58)
  30 min: number analyzed (Participants) | 32 | 25
  30 min | 90.78 (15.50) | 87.24 (21.02)
  60 min: number analyzed (Participants) | 32 | 25
  60 min | 90.03 (14.25) | 84.04 (14.34)
  240 min: number analyzed (Participants) | 32 | 25
  240 min | 91.22 (14.45) | 82.40 (17.92)

3. Secondary Outcome: Patient Vital Signs - Respiratory Rate [RR]
Description: Respiratory rate, measured in breaths per minute (brpm)
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients who had their Respiratory Rate collected during the four different timepoints in the study.
Measure: Mean (Standard Deviation); unit: Breaths per min
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
Breaths per min
  Baseline | 20.9 (5.00) | 21.2 (6.09)
  30 min: number analyzed (Participants) | 32 | 25
  30 min | 21.13 (6.41) | 22.12 (6.90)
  60 min: number analyzed (Participants) | 32 | 25
  60 min | 20.56 (5.30) | 21.32 (7.05)
  240 min: number analyzed (Participants) | 32 | 25
  240 min | 20.97 (4.82) | 20.92 (6.30)

4. Secondary Outcome: Patient Vital Signs - Oxygen Saturation [SpO2]
Description: SpO2 measured as percentage of oxygen saturation (%)
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients who had their SPO2 collected during the four timepoints in the study.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
percentage of oxygen saturation
  Baseline | 94.4 (7.42) | 96.8 (3.37)
  30 min: number analyzed (Participants) | 32 | 25
  30 min | 95.69 (3.46) | 96.80 (3.89)
  60 min: number analyzed (Participants) | 32 | 25
  60 min | 95.78 (3.08) | 97.28 (3.29)
  240 min: number analyzed (Participants) | 32 | 25
  240 min | 95.56 (2.91) | 97.16 (3.44)

5. Secondary Outcome: Patient Communication Capability - Patient Stability Index
Description: Patient stability index, measured by patient's ability to speak in full sentences, rated on a 0-100 scale. Higher scores indicate a better outcome.
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients that had the Stability Index collected during the four time points in the study.
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
units on a scale (0-100)
  Baseline | 62.00 (28.00) | 62.50 (23.09)
  30 min: number analyzed (Participants) | 32 | 25
  30 min | 73.81 (18.79) | 68.92 (17.23)
  60 min: number analyzed (Participants) | 32 | 25
  60 min | 77.75 (17.97) | 76.48 (15.78)
  240 min: number analyzed (Participants) | 32 | 25
  240 min | 82.28 (17.67) | 82.00 (19.37)

6. Secondary Outcome: Patient Venous Blood Gas - pH
Description: pH, measured as units on a pH scale from 0 - 14. Neutral scores indicate a better outcome.
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients that had this lab value collected during the four time points in the study.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
pH
  Baseline | 7.27 (.06) | 7.27 (.04)
  30 min: number analyzed (Participants) | 31 | 25
  30 min | 7.3 (.06) | 7.28 (0.06)
  60 min: number analyzed (Participants) | 31 | 25
  60 min | 7.31 (0.06) | 7.3 (0.07)
  240 min: number analyzed (Participants) | 31 | 25
  240 min | 7.31 (0.06) | 7.31 (0.06)

7. Secondary Outcome: Patient Venous Blood Gas - Venous PCO2
Description: Partial pressure of CO2 (PCO2), measured in mmHg
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients that had PCO2 collected during the four time points during the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
mmHg
  Baseline | 77.8 (13.6) | 76.5 (13.6)
  30 min: number analyzed (Participants) | 31 | 25
  30 min | 72.56 (15.71) | 73.22 (19.04)
  60 min: number analyzed (Participants) | 31 | 25
  60 min | 71.19 (14.85) | 70.95 (19.56)
  240 min: number analyzed (Participants) | 31 | 25
  240 min | 68.76 (13.68) | 67.29 (20.03)

8. Secondary Outcome: Patient Basic Metabolic Panel - Sodium
Description: Sodium [Na+], measured in mEq/L
Time Frame: Baseline, at study start only
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
mEq/L | 139.9 (3.5) | 140.4 (3.1)

9. Secondary Outcome: Patient Basic Metabolic Panel - Potassium
Description: Potassium [K+], measured in mEq/L
Time Frame: Baseline, at study start only
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
mEq/L | 4.4 (.63) | 4.4 (.66)

10. Secondary Outcome: Patient Basic Metabolic Panel - Chloride
Description: Chloride [Cl-], measured in mEq/L
Time Frame: Baseline, at study start only
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
mEq/L | 97.7 (6.4) | 99.9 (5.3)

11. Secondary Outcome: Patient Basic Metabolic Panel - Lactate
Description: Lactate, measured in mEq/L
Time Frame: Baseline, at study start only
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
mEq/L | 1.6 (1.25) | 1.2 (.84)

12. Secondary Outcome: Patient Basic Metabolic Panel - Glucose
Description: Glucose, measured in mg/dL
Time Frame: Baseline, at study start only
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
mg/dL | 133.8 (54.83) | 137.2 (40.03)

13. Secondary Outcome: Patient Base Excess - Base Excess
Description: Base Excess, measured in mEq/L
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients that had this lab value collected at the timepoints during the study.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 23 | 23
mEq/L
  Baseline | 6.7 (4.91) | 7.7 (5.56)
  30 min: number analyzed (Participants) | 18 | 16
  30 min | 7.43 (4.52) | 7.74 (7.03)
  60 min: number analyzed (Participants) | 18 | 16
  60 min | 6.71 (4.50) | 7.48 (6.45)
  240 min: number analyzed (Participants) | 18 | 16
  240 min | 5.97 (5.50) | 6.39 (6.74)

14. Secondary Outcome: Patient Bicarbonate - Bicarbonate
Description: Bicarbonate, measured in mEq/L
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients that had this lab value collected during the four time points in the study.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 33 | 32
mEq/L
  Baseline | 32.0 (7.63) | 33.8 (6.60)
  30 min: number analyzed (Participants) | 32 | 26
  30 min | 33.18 (5.61) | 32.43 (9.86)
  60 min: number analyzed (Participants) | 32 | 26
  60 min | 32.75 (5.69) | 32.45 (8.11)
  240 min: number analyzed (Participants) | 30 | 26
  240 min | 30.93 (8.73) | 32.18 (7.35)

15. Other Pre Specified Outcome: Patient Perception Score - Relief of Symptoms
Description: Patient's subjective assessment of relief of their symptoms while on therapy, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients that had this data collected at the four time points during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
units on a scale
  Baseline | 34.8 (24.81) | 38.5 (22.19)
  30 min: number analyzed (Participants) | 31 | 24
  30 min | 28.45 (22.26) | 38.05 (19.91)
  60 min: number analyzed (Participants) | 31 | 24
  60 min | 24.68 (19.86) | 27.82 (20.10)
  240 min: number analyzed (Participants) | 31 | 24
  240 min | 28.48 (24.09) | 24.58 (21.80)

16. Other Pre Specified Outcome: Patient Perception Score - Comfort/Tolerance
Description: Patient's subjective assessment of their comfort and tolerance of therapy during the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: During four time points in the study over the course of four hours; Baseline, 30 min, 60 min, and 240 min
Population: Patients who had their score collected during the four different timepoints in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 36 | 32
units on a scale
  Baseline | 34.8 (24.81) | 38.5 (22.19)
  30 min: number analyzed (Participants) | 31 | 22
  30 min | 28.39 (22.53) | 44.82 (24.41)
  60 min: number analyzed (Participants) | 31 | 22
  60 min | 22.35 (19.49) | 42.41 (28.30)
  240 min: number analyzed (Participants) | 31 | 24
  240 min | 20.13 (23.45) | 43.25 (32.02)

17. Other Pre Specified Outcome: Clinician Perception Score - Expected/Perceived Outcomes
Description: Clinician's subjective assessment of the expected and perceived patient outcomes as a result of therapy following testing, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: At study end, 4 hours from study start
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 31 | 25
units on a scale | 23.26 (14.33) | 16.32 (14.52)

18. Other Pre Specified Outcome: Clinician Perception Score - Patient Comfort/Tolerance
Description: Clinician's subjective assessment of the patient's comfort and tolerance of therapy during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: At study end, 4 hours from study start
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 31 | 25
units on a scale | 17.58 (13.61) | 22.04 (20.87)

19. Other Pre Specified Outcome: Clinician Perception Score - Ease of Use
Description: Clinician's subjective assessment of the ease of use of therapy during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: At study end, 4 hours from study start
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 31 | 25
units on a scale | 16.45 (16.25) | 15.08 (18.68)

ADVERSE EVENTS:
Time Frame: Over the course of the study, which took place for a total of 4 hours.
Description: The investigator will determine whether any adverse events have occurred. If any adverse event occurs, either anticipated or unanticipated, the investigators will immediately contact the sponsor representative (site monitor) which is indicated on the fist page of the protocol. The case report forms will have a list of predetermined adverse events to be used actively to screen during the study procedures.
Arm/Group | High Velocity Nasal Insufflation (HVNI) | Noninvasive Positive Pressure Ventilation (NIPPV)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 0/36 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04709562/Prot_SAP_000.pdf